CLINICAL TRIAL: NCT00760266
Title: An 8-week Randomized, Double-blind, Parallel-group, Multi-center, Active-controlled Dose Escalation Study to Evaluate the Efficacy and Safety of Aliskiren HCTZ (300/25 mg) Compared to HCTZ (25 mg) in Older Patients With Stage 2 Systolic Hypertension
Brief Title: Blood Pressure Lowering of Aliskiren HCTZ Compared to HCTZ in Stage 2 Systolic Hypertension in Older Population
Acronym: ACTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPP100A2411
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Results first posted 2011-01-21 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
Keywords: Hypertension; older population; aliskiren; hydrochlorothiazide; systolic blood pressure; diastolic blood pressure; amlodipine, stage 2
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren/HCTZ 300/25 mg (Experimental)
  Interventions: Drug: Aliskiren
- HCTZ 25 mg (Active Comparator)
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 150 mg for 1 week, Aliskiren 300 mg (with or without amlodipine)for 7 weeks
  Arms: Aliskiren/HCTZ 300/25 mg
Drug: Hydrochlorothiazide — Hydrochlorothiazide (HCTZ) 12.5 mg for week 1; Hydrochlorothiazide (HCTZ) 25 mg (with or without amlodipine)for 7 weeks
  Arms: HCTZ 25 mg

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of initial use of a fixed dose combination of aliskiren Hydrochlorothiazide (HCTZ) compared to Hydrochlorothiazide in older population with Stage 2 systolic hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients, ≥ 55 years old
2. Patients with essential hypertension
3. Prior to randomization: Patients must have an office cuff mean sitting Systolic Blood Pressure ≥ 160 mm Hg and < 200 mm Hg
4. Patients who are eligible and able to participate in the study, and who are willing to give informed consent before any assessment is performed

Exclusion Criteria:

1. Office blood pressure measured by cuff (msSBP ≥ 200 mm Hg and/or msDBP ≥ 110 mm Hg) at Visits 1-5
2. History or evidence of a secondary hypertension of any etiology (e.g., uncorrected renal artery stenosis, pheochromocytoma).
3. History of hypertensive encephalopathy or heart failure (New York Heart Association [NYHA] Class II-IV)
4. Cerebrovascular accident, transient ischemic cerebral attack (TIA), myocardial infarction, coronary bypass surgery, or any percutaneous coronary intervention (PCI) within 1 year prior to Visit 1
5. Serum sodium less than the lower limit of normal, serum potassium < 3.5 mEq/L (corresponding to 3.5 mmol/L) or ≥ 5.3 mEq/L (corresponding to 5.3 mmol/L), or dehydration at Visit 1.
6. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL)
7. Use of other investigational drugs within 30 days of enrollment.

Other exclusions may apply.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2008-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sites in USA, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Yan JH, Jarugula V, Sabo R, Papst CC, Zhang J, Dole WP. Pharmacokinetics and pharmacodynamics of aliskiren/hydrochlorothiazide single-pill combination tablets and free combination of aliskiren and hydrochlorothiazide. J Clin Pharmacol. 2012 May;52(5):645-55. doi: 10.1177/0091270011405499. Epub 2011 Jun 9. PMID 21659626

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren/HCTZ: Aliskiren / Hydrochlorothiazide (HCTZ) 150/12.5 mg: 1 week, Aliskiren / HCTZ 300/25 mg (with or without amlodipine): 7 weeks
- HCTZ: Hydrochlorothiazide (HCTZ) 12.5 mg: 1 week, HCTZ 25 mg (with or without amlodipine): 7 weeks
Period: Overall Study
Arm/Group | Aliskiren/HCTZ | HCTZ
Started | 228 | 223
Completed | 204 | 205
Not Completed | 24 | 18
Not completed — Adverse Event | 13 | 7
Not completed — Abnormal laboratory value(s) | 1 | 0
Not completed — Abnormal test procedure result(s) | 1 | 0
Not completed — Lack of Efficacy | 2 | 2
Not completed — Protocol deviation | 2 | 4
Not completed — Patient withdrew consent | 3 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Administrative Problems | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren/HCTZ | HCTZ | Total
Number analyzed (Participants) | 228 | 223 | 451
Age Continuous [Mean (Standard Deviation); unit: years] | 64.5 (7.57) | 65.1 (6.96) | 64.8 (7.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 100 | 227
  Male | 101 | 123 | 224

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) From Baseline to Week 4
Time Frame: Baseline and Week 4
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren/HCTZ | HCTZ
Number analyzed (Participants) | 225 | 222
mm Hg | -29.6 (1.0) | -22.3 (1.0)

2. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) From Baseline to Week 4
Time Frame: Baseline and Week 4
Population: Full analysis set, restricted to baseline msDBP >= 90 mmHg
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren/HCTZ | HCTZ
Number analyzed (Participants) | 130 | 133
mm Hg | -11.1 (0.8) | -9.2 (0.8)

3. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) and Mean Sitting Diastolic Blood Pressure (msDBP) (in Patients With msDBP ≥90 mmHg at Baseline) From Baseline to Week 8
Time Frame: Baseline and Week 8
Population: Full analysis set, restricted for msDBP to those with baseline msDBP at least 90 mm Hg)
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren/HCTZ | HCTZ
Number analyzed (Participants) | 225 | 222
mm Hg
  msSBP | -33.2 (1.0) | -25.7 (1.0)
  msDBP (N = 130 , 133) | -13.3 (0.8) | -10.1 (0.8)

4. Secondary Outcome: Percentage of Responders at Week 4 and Week 8
Description: Responders defined as mean sitting Systolic Blood Pressure < 140 mmHg or reduction of ≥ 20 mmHg from baseline
Time Frame: At 4 weeks and 8 weeks
Population: Full analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Aliskiren/HCTZ | HCTZ
Number analyzed (Participants) | 225 | 222
Percentage of Participants
  Week 4 | 73.3 | 55.9
  Week 8 | 83.1 | 67.6

5. Secondary Outcome: Percentage of Subjects Achieving Blood Pressure Control at Weeks 4 and 8
Description: Blood pressure control defined as mean sitting Systolic Blood Pressure < 140 mm Hg and mean sitting Diastolic Blood Pressure < 90 mm Hg
Time Frame: At Weeks 4 and 8
Population: Full analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Aliskiren/HCTZ | HCTZ
Number analyzed (Participants) | 225 | 222
Percentage of Participants
  week 4 | 49.8 | 33.3
  week 8 | 62.2 | 39.2

ADVERSE EVENTS:
Description: One patient was excluded from this analysis as he/she was inadvertently randomized into the study but did not receive study drug.
Groups:
- Aliskiren / HCTZ: Aliskiren HCTZ 150/12.5 mg: 1 week, Aliskiren HCTZ 300/25 mg (with or without amlodipine): 7 weeks
- HCTZ: HCTZ 12.5 mg: 1 week, HCTZ 25 mg (with or without amlodipine): 7 weeks
Arm/Group | Aliskiren / HCTZ | HCTZ
Serious Adverse Events (participants affected / at risk) | 4/227 | 3/223
Other Adverse Events (participants affected / at risk) | 17/227 | 26/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren / HCTZ (N=227) | HCTZ (N=223)
Colitis (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Renal function test abnormal (Investigations) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren / HCTZ (N=227) | HCTZ (N=223)
Dizziness (Nervous system disorders) | 13 | 9
Headache (Nervous system disorders) | 4 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.